CLINICAL TRIAL: NCT02574208
Title: Acceptability and Feasibility of HIV Testing by ELISA or Rapid Test to Adult Patients Consulting Their General Practitioner in Paris, France: A Multi-center Prospective Randomized Study
Brief Title: Acceptability/Feasibility of HIV Testing by ELISA or Rapid Test to Adult Patients in Paris, France
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hopital Lariboisière (Other)
Responsible Party: Principal Investigator, Célia Lloret-Linares, MD PhD, MD PhD, Hopital Lariboisière
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: DEPICAB
Record Dates: First submitted 2015-09-30; First posted 2015-10-12 (Estimated); Last update posted 2016-11-22 (Estimated); Status verified 2016-11

CONDITIONS: HIV
Keywords: Adult outpatients; Paris, France

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- "HIV testing by ELISA" (Active Comparator): Patients enrolled in this arm will be tested by usual HIV Elisa
  Interventions: Procedure: HIV testing by ELISA
- "HIV testing by rapid test" (Experimental): Patients enrolled in this arm will be tested by the new rapid HIV test
  Interventions: Procedure: HIV testing by rapid test

INTERVENTIONS:
Procedure: HIV testing by ELISA — HIV testing randomized between ELISA or rapid test
  Arms: "HIV testing by ELISA"
Procedure: HIV testing by rapid test — HIV testing randomized between ELISA or rapid test
  Arms: "HIV testing by rapid test"

SUMMARY:
CDC recommends universal HIV testing in all adults, at least once during life, to reduce the pool of infected patients unaware of their status. Routine universal HIV testing can use "classical" ELISA tests from serum, or rapid tests, ideally from finger-stick whole blood (FSB), which have shown close predictive values from classical tests. The investigators will compare the acceptability and feasibility of the two methods.

DETAILED DESCRIPTION:
The multi-center prospective randomized study will compare the acceptability and feasibility of routine universal HIV testing to adult patients consulting their general practitioner in Paris, France, using either the " classical " ELISA tests from serum or rapid tests from FSB (Insti®).

ELIGIBILITY:
Inclusion Criteria:

* adult patients consulting their general practitioner in Paris, France

Exclusion Criteria:

* patients previously known as HIV-positive,
* patients who declare having been tested HIV-negative less than three months ago,
* patients who can not give informed consent

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 260 (Actual)
Dates: Start 2015-10; Primary Completion 2015-12 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
acceptability of HIV testing | immediately after HIV testing proposal
  answer by "yes" or "no" to the single following question: "do you agree to perform an HIV test?"

SECONDARY OUTCOMES:
feasibility of HIV testing | one month after HIV testing proposal
  Number of HIV test results recovered within a month upon enrollment

CONTACTS AND LOCATIONS:
Overall Officials: Pierre O Sellier, M.D., Ph.D., Principal Investigator — Hopital Lariboisiere

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Prost A, Griffiths CJ, Anderson J, Wight D, Hart GJ. Feasibility and acceptability of offering rapid HIV tests to patients registering with primary care in London (UK): a pilot study. Sex Transm Infect. 2009 Sep;85(5):326-9. doi: 10.1136/sti.2008.033233. Epub 2009 May 31. PMID 19487214